CLINICAL TRIAL: NCT04367077
Title: A Phase 2/3 Study to Assess the Safety and Efficacy of MultiStem® Therapy in Subjects With Acute Respiratory Distress Syndrome (ARDS) Due to Coronavirus Disease (COVID-19)
Brief Title: MultiStem Administration for COVID-19 Induced ARDS (MACoVIA)
Acronym: MACoVIA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healios K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B04-03
Record Dates: First submitted 2020-04-27; First posted 2020-04-29 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: ARDS
Keywords: COVID19; respiratory distress; adult stem cells
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MultiStem (Experimental)
  Interventions: Biological: MultiStem
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: MultiStem — intravenous infusion
  Arms: MultiStem
Biological: Placebo — intravenous infusion
  Arms: Placebo

SUMMARY:
Multicenter investigation featuring an open-label lead-in followed by a double blinded, randomized, placebo-controlled Phase 2/3 part to evaluate the safety and efficacy of MultiStem therapy in subjects with moderate to severe Acute Respiratory Distress Syndrome (ARDS) due to pathogens including COVID-19.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of new acute-onset moderate to severe ARDS, as defined by the Berlin criteria, requiring an endotracheal or tracheal tube, Evidence of pneumonia or severe localized or systemic infection

Exclusion Criteria:

Moribund subject who, in the opinion of the Investigator, is not expected to survive at least 48 hours and End-stage severe chronic lung disease

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Ventilator-Free Days | Day 0 through Day 28.
Safety and Tolerability as measured by the incidence of treatment-emergent adverse events as assessed by CTCAE v5.0. | Day 28

SECONDARY OUTCOMES:
All-cause mortality | Day 60
Ranked hierarchical composite outcome of alive and ventilator-free | Day 28
Ventilator-free days | Day 0 through Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jenkins, MD, Study Director — Healios K.K.
Locations (4):
- United States (4):
  - Athersys Investigational Site 107, Chicago, Illinois
  - Athersys Investigational Site 103, Akron, Ohio
  - Athersys Investigational Site 101, Cleveland, Ohio
  - Athersys Investigational Site 102, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No